CLINICAL TRIAL: NCT03423589
Title: Modulation of Type 1 Diabetes Susceptibility Through VSL#3 Probiotic-induced Alterations in the Intestinal Microbiota
Brief Title: Modulation of Type 1 Diabetes Susceptibility Through the Use of Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, MD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1171017
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Type1diabetes; Type1 Diabetes Mellitus
Keywords: Siblings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VSL#3 (Experimental): Participants will be given the probiotic supplement VSL#3, a commercially available product. VSL#3 is taken by mouth, either once or twice daily, and is dispensed in sachets, each containing 450 billion colony forming units of bacterial strains. Participants will undergo a screening visit. They will be asked to provide a stool sample by the next visit. Within 3 weeks they will return with a stool sample and receive the VSL#3 sachets as well as another stool collection kit. After 6 weeks of taking VSL#3, they will return for their final visit, with their stool sample. Blood will be drawn at the second and third visits.
  Interventions: Dietary Supplement: VSL#3

INTERVENTIONS:
Dietary Supplement: VSL#3 — VSL#3 is a commercially available probiotic supplement manufactured and distributed by Alfasigma USA, Inc of Covington, Louisiana, USA. As with other probiotics, VSL#3 is considered a supplement and is not FDA-approved or regulated. VSL#3 contains eight probiotic strains: bifidobacteria (B. longum, B. infantis, and B. breve), lactobacilli (L. acidophilus, L. casei, L. bulgaricus, and L. plantarum) and Strepococcus thermophiles.

SUMMARY:
Investigators aim to further the understanding of environmental factors that underlie the progression to Type 1 diabetes (T1D). Dysbiosis, defined as alterations in intestinal microbiota composition and function, has been hypothesized to increase the risk of developing T1D in those with genetic susceptibility. Dysbiosis may result from modern dietary habits, such as broad consumption of the highly processed Western Diet, or by widespread use of antibiotics. Here, investigators propose to examine the impact of dysbiosis on the endogenous innate inflammation known to exist within families affected by T1D and if probiotic supplementation may beneficially modulate this inflammatory state.

Participants will be asked to take the probiotic VSL#3 daily for six weeks. Stool and blood samples will be analyzed before and after the six week course of probiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 5-17 years of age
2. Full-sibling of an individual with a clinical diagnosis of Type 1 diabetes
3. Treatment naïve of any immunomodulatory agent
4. Naïve of any probiotic supplement within the past 12 months

Exclusion Criteria:

1. Presence of severe/active disease that interferes with dietary intake
2. Chronic use of medications known to affect gastrointestinal function, such as stool softeners or laxatives
3. Diagnosis of celiac disease and/or following a gluten-free diet
4. Presence of significant and sustained gastrointestinal symptoms within the prior 6 weeks (e.g., severe abdominal pain, worsening constipation, diarrhea, or recurrent nausea +/- vomiting)
5. Chronic inflammatory or autoimmune disease with the exception of well-controlled hypothyroidism or intermittent or mild persistent asthma not requiring the use of daily inhaled steroids
6. Use of any medications that could affect intestinal microbiota within the previous 3 months (e.g., antibiotics, prebiotics, or probiotics)
7. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results
8. Female participants of child-bearing age must not be pregnant

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Alterations in Plasma-Induced Transcriptional Analysis | 2 years (study duration)
  Examine the probiotic-induced alterations in the plasma-induced transcriptional analysis

SECONDARY OUTCOMES:
Intestinal Microbiota | 2 years (study duration)
  Examine the intestinal microbiota, plasma microbial antigen levels as a marker of gut barrier function

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided